CLINICAL TRIAL: NCT01377532
Title: Compassionate Use of 131I-MIBG for Patients With Malignant Pheochromocytoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CompUse MIBG Pheo
Record Dates: First submitted 2011-06-13; First posted 2011-06-21 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Pheochromocytoma; Paraganglioma; MIBG; 131I-MIBG; Resistant; Relapsed; Treatment; UCSF; Pediatric; Adult; Oncology
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Recurrence; Neoplasms | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: 131 I-Metaiodobenzylguanidine (131 I-MIBG) — Therapeutic 131I-MIBG will be synthesized at Nuclear Diagnostic Products (NDP; Rockaway, New Jersey) with specific activities of 9-18 Ci/mmole. The therapeutic dose: 8-12 mCi/kg (maximum 500 mCi ± 10% at investigator's discretion) will be diluted in 25 ml of normal saline, and will be infused intravenously through a patient's peripheral or central line over 120 minutes. The patient will remain in a radiation protected isolation room until radiation emissions are ≤ 2 mr/hr at a 1 meter distance or meets institutional and state guidelines. This usually takes 4-6 days. In all cases, special shielding will be equipped in the room to minimize exposure to the outside environment and personnel will observe institutional radiation safety precautions. A radiation safety officer will instruct the patient, family, and caretakers about specific UCSF radiation safety guidelines for both hospitalization and discharge.
  Other Names: 131I-MIBG

SUMMARY:
This is a compassionate use protocol to allow palliative therapy for patients with malignant pheochromocytoma and paragangliomas.

DETAILED DESCRIPTION:
Pheochromocytomas (PHEO) and paragangliomas (PGL) are rare tumors, with an incidence of 2-8 cases per million annually. These tumors develop in both children and adults. About 15-20% metastasize. Chemotherapy for this tumor usually consists of a combination of cyclophosphamide, vincristine, and dacarbazine delivered over two days and repeated every 3 weeks. Such combined chemotherapy is ineffective for the majority of patients with metastatic PHEO/PGL. A few patients with malignant PHEO have experienced remissions with sunitinib, but the drug may produce severe toxicity and the experience with that drug is limited. Those patients who do experience a remission with chemotherapy must continue it indefinitely to stay in remission. However, most such patients experience such severe side effects from the chemotherapy (marrow suppression, neuropathy, etc) that their chemotherapy must be discontinued. Thus, chemotherapy is either ineffective or intolerable for the vast majority of patients with metastatic PHEO/PGL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Refractory or relapsed PHEO/PGL with original diagnosis based on tumor histopathology or the finding of PHEO/PGL tumor cells in the bone marrow. The diagnosis may also be based upon the presence of high plasma fractionated metanephrines or high urine catecholamines/metanephrines with diagnostic MIBG uptake.
* Age: > 2 years and able to cooperate with radiation safety restrictions during therapy period.
* Disease status: It must be determined that either the PHEO/PGL tumors are not amenable to safe surgical resection or are metastatic. Disease evaluable by MIBG scan must be present within 6 weeks of study entry and subsequent to any intervening therapy.
* Life Expectancy: greater than 3 months.
* Lanksy and Karnofsky Performance Status: 70% or higher.
* Prior Therapy: Patients may enter this study with or without having had other therapy for recurrent tumor. Patients may be treated who have not had chemotherapy or radiation therapy. Patients may also be treated who have failed to respond to standard chemotherapy or radiation therapy. Patients must have fully recovered from the toxic effects of any prior therapy. At least 2 weeks should have elapsed since any anti-tumor therapy and the patient must meet hematologic criteria below. Three months should have elapsed in the case of completing radiation to any of the following fields: total craniospinal, total abdominal, whole lung, total body irradiation). Cytokine therapy (eg G-CSF, GM-CSF, IL-6, erythropoietin) must be discontinued a minimum of 24 hours prior to MIBG therapy. Prior 131I-MIBG therapy is allowed if > 8 weeks from previous treatment. Cumulative lifetime dose of 131I-MIBG, including the planned treatment, should not exceed 36 mCi/kg.
* Liver function: bilirubin < 2x upper limit of normal (ULN). Exception: Gilbert syndrome); AST < 10x ULN.
* Kidney function: Creatinine =< 2x ULN.
* Hematopoietic Criteria Patients must have adequate hematopoietic function (without transfusion): ANC >750 x 10E9/L; Platelets >50 x 10E9/L if stem cells are not available; if stem cells are available, the patient should be independent of platelet transfusions with a platelet count of at least 20 x 10E9/L. Hemoglobin >10g/dl at time of treatment (transfusion allowed). Patients with granulocytopenia and/or thrombocytopenia due to tumor metastatic to the bone marrow may be eligible after discussion with Dr. Fitzgerald or designee.
* Normal lung function as manifested by no dyspnea at rest or exercise intolerance, no oxygen requirement.
* No clinically significant cardiac dysfunction, normal EKG and EJ >50%

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand therapy. Any significant organ impairment should be discussed with the Study Chair or Vice Chair prior to patient entry.
* Patients with proteinuria in the absence of urinary infection 4 weeks prior to the planned treatment date.
* Because of the teratogenic potential of the study medications, no patients who are pregnant or breast feeding will be allowed. Patients of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible pregnancy.
* Patients who are on hemodialysis.
* Patients with active infections that meet grade 3-4 toxicity criteria.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fitzgerald, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States